CLINICAL TRIAL: NCT04557423
Title: Evidence-Based Approach to Empower Asian American Women in Cervical Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Carolyn Fang, PhD, Professor, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-1058
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evidence-Based Intervention (Active Comparator): Culturally appropriate educational intervention focused on cervical cancer screening, with navigation assistance provided.
  Interventions: Behavioral: Community-Based Education; Behavioral: Navigation to Screening
- HPV Self-Sampling (Experimental): Previously tested evidence-based intervention (i.e. culturally appropriate educational intervention focused on cervical cancer screening, with navigation assistance provided). Participants will also receive a self-sampling kit.
  Interventions: Behavioral: Community-Based Education; Behavioral: Navigation to Screening; Behavioral: HPV Self-Sampling

INTERVENTIONS:
Behavioral: Community-Based Education — A previously evaluated educational intervention delivered in community settings. Includes culturally- and linguistically-appropriate materials.
Behavioral: Navigation to Screening — Community health educators provide navigation assistance to access clinic-based cervical cancer screening.
Behavioral: HPV Self-Sampling — An HPV self-sampling kit will be provided for home-based collection of cervical samples. Samples will be sent for analysis of HPV subtypes.
  Arms: HPV Self-Sampling

SUMMARY:
This is a randomized trial to evaluate the effects of a community-based intervention on increasing cervical cancer screening rates in underserved Asian American (Korean, Vietnamese, and Chinese) women. All women will receive an educational program and navigation assistance. Women in the intervention condition will also receive a self-sampling kit for self-collection of a cervical sample for HPV testing. The investigators will evaluate whether the inclusion of a self-sampling kit increases the proportion of Asian American women who participate in cervical cancer screening.

DETAILED DESCRIPTION:
Aim 1: Compare rates of providing a self-collected sample vs. obtaining clinic-based screening among 1100 Asian American women. It is hypothesized that the proportion of women in the HPV self-sampling program who provide a self-collected sample will be higher than the proportion of women in the clinic-based program who obtain clinic-based screening.

Aim 2: Examine mediators of participation. The investigators will examine both individual- and social/environmental-level factors associated with participation across both programs. It is hypothesized that higher levels of perceived self-efficacy, lower levels of embarrassment, and fewer barriers will be associated with higher rates of participation in both conditions. Further, it is hypothesized that women in the HPV self-sampling program will report greater self-efficacy, less embarrassment, and fewer barriers compared to women in the clinic-based program.

Aim 3: Assess the relative cost-effectiveness of HPV self-sampling vs. clinic-based screening. The investigators will conduct an incremental cost-effectiveness analysis from a societal perspective incorporating trial-based direct medical and participant-borne costs associated with HPV self-sampling vs. clinic-based screening. It is hypothesized that the self-sampling program will be less costly to implement and achieve a higher participation rate.

ELIGIBILITY:
Inclusion Criteria:

* Women who are of Asian race and self-identify as Korean, Vietnamese, or Chinese
* are 30-65 years of age
* are overdue for cervical cancer screening (e.g., no cytology-based screening within the past 3 years; no hrHPV testing either alone or in combination with cytology in the past 5 years)

Exclusion Criteria:

* have a prior diagnosis of cervical cancer or cervical abnormality (e.g., dysplasia)
* had a hysterectomy with removal of the cervix
* have a compromised immune system (e.g., known HIV)
* unable to provide informed consent

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Participation in screening | 6 months
  The number of women who obtain clinic-based screening or return a self-collected sample

SECONDARY OUTCOMES:
Program delivery cost | 6 months
  The costs associated with delivering each program. This will include: (1) Participant costs (time spent participating in educational sessions and time required to complete screening; transportation costs, if incurred); (2) Screening costs (cost of clinic-based screening, or cost of the HPV self-sampling kit); (3) Program delivery costs (community health educator time for conducting the educational programs, time will be valued at wage rates including benefits; costs of educational materials [flyers, booklets] and reminder letters); (4) Navigation costs (time and labor involved in navigating women to the clinic for screening will be documented using a log of CHE time and expenses incurred).

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Temple University Lewis Katz School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data and associated documentation can be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. All procedures will be compliant with NIH regulations on the distribution of unique research resources.